CLINICAL TRIAL: NCT05901324
Title: Efficacy of Lenalidomide Maintenance in Primary Central Nervous System Lymphoma and Primary Vitreoretinal Lymphoma
Brief Title: Efficacy of Lenalidomide Maintenance in Primary Central Nervous System Lymphoma and Primary Vitreoretinal Lymphoma: a Phase II, Open-label, Single-arm Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Attending Physician, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202303123MIPA
Record Dates: First submitted 2023-06-04; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Primary Central Nervous System Lymphoma and Primary Vitreoretinal Lymphoma
Keywords: primary central nervous system lymphoma and primary vitreoretinal lymphoma; primary vitreoretinal lymphoma
MeSH Terms: interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maintenance therapy with lenalidomide as the maintenance therapy for patients with PCNSL or PVRL (Experimental)
  Interventions: Radiation: intensity-modulated radiotherapy (IMRT)

INTERVENTIONS:
Radiation: intensity-modulated radiotherapy (IMRT) — 1.8 Gy of 4-6 MV X-ray to a total dose of 23.4 Gy (13 fractions) will be delivered.

SUMMARY:
Therefore, we intend to conduct a phase II study to evaluate the efficacy of maintenance therapy with lenalidomide as the maintenance therapy for patients with PCNSL or PVRL who have achieved CR or partial response after HD-MTX-based induction therapy followed by reduced-dose WBRT.Twentypatients with PCNSL or PVRL will be recruited. The primary outcome is 2-year progression-free survival from the first date of reduced-dose WBRT. Besides, the safety and the incidence of cute and late neurotoxicity related to reduced-dose WBRT, the single nucleotide polymorphism assay,and the clinical applications of plasma and CSF circulating tumor DNA and CSF lactate level will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Those who have been diagnosed with histopathological- or CSF/vitreous fluid flow cytometry- confirmedPCNSL/PVRL, DLBCL subtype and who are above 18 years of age.
2. Those who have completed standard HD-MTX-based remission induction chemotherapy followed by reduced-dose WBRT and reached a CR or PR
3. Patients must be able to tolerate MRI scans and lumbar punctures and/or Ommaya taps.
4. With sufficient organ and bone marrow function, and no severe hematopoietic, heart, lung, liver, kidney, thyroid dysfunction, and immune deficiency
5. ECOG PS 0-2
6. Those who can take oral medication
7. Written informed consent under institutional guidelines.
8. Female patients of child-bearing potential (FCBP) must have two negative pregnancy tests (sensitivity of at least 25 mIU/mL) prior to starting lenalidomide. The first pregnancy test must be performed within 10 to 14 days prior to the start of lenalidomide, and the second pregnancy test must be performed within 24 hours prior to the start of lenalidomide
9. Effective method of contraception should be used during and for 28 days following the last dose of the drug
10. Male patients must use an effective barrier method of contraception during study and 28 days following the last dose if sexually active with a FCBP

Exclusion Criteria:

1. Patients who are planned to undergo auto-SCT after induction chemotherapy
2. Disease involving extra-CNSat the time of initial diagnosis
3. Previous treatment with lenalidomide or WBRT
4. Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within six months prior to 1st day of 1st cycle
5. Acute active infection requiring systemic antibiotics, antiviral (except antiviral therapy directed at hepatitis B) or antifungal agents
6. Known human immunodeficiency (HIV) seropositive
7. Those who are unable to take oral medication or unable to take antiplatelet therapy for the purpose of thromboembolism prevention.
8. Patients with a history of malignant tumors other than the target diseases except for the following cases oIf the tumor has not been treated for at least 5 years or is disease-free oPatients at least 1 year after complete resection of basal cell carcinoma / squamous cell carcinoma or successful treatment of cervical epithelial cancer
9. Adverse reactions within 30 days prior to screening Severe gastrointestinal bleeding exceeding Grade 2 according to the Common Terms Criteria 4.03 version criteria
10. Occurrence of blood clots or embolism within 6 months before starting screening
11. Patients with hypersensitivity to THIS DRUG and other ingredients of THIS DRUG (e.g., angioedema, Stevens-Jones syndrome, toxic epidermal necrosis, etc.)
12. Female patients who are pregnant or lactating
13. The Patient is unwell or unable to participate in all required study evaluations and procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2031-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of tumor progression or death from all causes from the starting date of reduced-dose WBRT to the end of maintenance therapy | 2-year

SECONDARY OUTCOMES:
The time from the starting date of reduced-dose WBRTto death from any cause. | 24months
The proportion of patients who achieve CR and PR. | 24months

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF